CLINICAL TRIAL: NCT02794805
Title: Evaluation of the Capability of the ¹³C-Octanoate Breath Test (OBT) Measurement to Differentiate Between Presence and Absence of HCC Determined by MRI in Patients With Chronic Liver Disease
Brief Title: Determination of HCC With Octanoate Breath Test vs. MRI Diagnosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HCC-MPBA-0514
Record Dates: First submitted 2016-06-05; First posted 2016-06-09 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCC positive (Experimental): Breath testing utilizing 13C is a safe, non-invasive means for measuring a certain pathway's metabolic rate. 13C is a stable, non-radioactive isotope which can be incorporated into a specific location within a test substrate so it would be released when the compound is metabolized by the liver. Hepatic metabolism of the compound is assessed by measuring the ratio of 13CO2/12CO2 in exhaled breath.
  Interventions: Device: ¹³C-Octanoate Breath Test
- HCC negative (Experimental): Breath testing utilizing 13C is a safe, non-invasive means for measuring a certain pathway's metabolic rate. 13C is a stable, non-radioactive isotope which can be incorporated into a specific location within a test substrate so it would be released when the compound is metabolized by the liver. Hepatic metabolism of the compound is assessed by measuring the ratio of 13CO2/12CO2 in exhaled breath.
  Interventions: Device: ¹³C-Octanoate Breath Test

INTERVENTIONS:
Device: ¹³C-Octanoate Breath Test — Octanoate Breath Test to be performed on subjects with suspected HCC
  Other Names: Caprylate; Sodium caprylate

SUMMARY:
An Octanoate breath test will be used to assess the presence of Hepatocellular Carcinoma in subjects with risk. The gold standard will be MRI.

DETAILED DESCRIPTION:
1. Informed consent will be obtained from all patients prior to enrollment.
2. The trial will be conducted in compliance with this protocol, with GCP standards, and the applicable regulatory requirements.
3. This study will be cross-sectional, where patients will be enrolled on a walk in basis. Once one arm is completed the other one will be enriched in order to obtain at least 50 positive and at least 50 negative HCC subjects as defined by MRI.
4. All patients will undergo AFP and US if they do not have results within the past three months.
5. If the patient undergoes liver FNA, the biopsy results will be evaluated for the presence of HCC.
6. For all patients, a case report form will be completed.
7. All patients will undergo a physical examination, and their medical history/concomitant medications, weight, height and age will be recorded. Furthermore, recent (past 3 months) blood test results, if available, may be recorded.
8. If relevant (woman of child bearing age), a pregnancy test will be performed to rule out pregnancy when performing the breath test.
9. All MRI negative patients with low OBT results will undergo additional MRI within 6 to 12 months post OBT to rule out HCC occurrence.
10. If available, all additional MRI/CT/US results will be recorded within the patient's CRF.

ELIGIBILITY:
Inclusion Criteria:

1. Any patients with chronic liver disease at risk for HCC.
2. Age ≥ 18 years.
3. Patient has an MRI result (positive or negative for HCC) up to 3 months prior to recruitment or will be scheduled for an MRI during the trial period.
4. Patient is naïve to HCC treatment (RFA or TACE or Oral HCC treatments) since last MRI.

Exclusion Criteria:

1. Any patients with chronic liver disease at risk for HCC.
2. Age ≥ 18 years.
3. Patient has an MRI result (positive or negative for HCC) up to 3 months prior to recruitment or will be scheduled for an MRI during the trial period.
4. Patient is naïve to HCC treatment (RFA or TACE or Oral HCC treatments) since last MRI.
5. Patients currently receiving total parenteral nutrition if they have contraindications to oral drugs.
6. Women who are pregnant or breast feeding.
7. Patient taking drugs that can interfere with octanoate metabolism or can also cause NAFLD independent of the metabolic syndrome, including: corticosteroids, amiodarone, tetracycline, valproic acid, methotrexate, stavudine, zidovudine.
8. Patient, based on the opinion of the investigator, should not be enrolled into this study.
9. Patient unable or unwilling to sign informed consent.
10. Patients that are participating in other clinical trials evaluating experimental treatments or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
13CO2/12CO2 ratio | 60 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - 302 Military Hopsital, Beijing
  - General Hospital of Beijing Military Region, Beijing

IPD SHARING:
Plan to Share IPD: No